CLINICAL TRIAL: NCT00029913
Title: A Multi-Site Evaluation of Virologic, Immunologic, and Clinical Natural History of Participants Enrolled in Phase I and Phase II HIV-1 Vaccine Protocols or HIV-1 Vaccine Preparedness Cohorts Who Develop HIV-1 Infection Subsequent to Trial Enrollment
Brief Title: A Study of Patients Who Develop HIV Infection After Enrolling in HIV Vaccine Trials or HIV Vaccine Preparedness Trials
Status: Completed | Type: Observational
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Erik Schwab, HVTN
Other Study IDs: HVTN 403; 5U01AI068614 (NIH)
Record Dates: First submitted 2002-01-24; First posted 2002-01-25 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: Placebos; AIDS Vaccines; CD4 Lymphocyte Count; Disease Progression; Viral Load; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Observation of participants includes a physical exam and collection of fluids. Study visits occur at Days 0, 7, 14, 28 and at Months 2, 3, 6 and every 6 months thereafter.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of participants who received HIV preventive vaccine and became infected.

SUMMARY:
Despite risk reduction counseling, some individuals in HIV vaccine trials or vaccine preparedness studies may engage in risk behavior that results in HIV infection. The purpose of the HVTN 403 study is to find out more about how persons respond to HIV infection if they have received an experimental HIV-1 vaccine before they became HIV infected.

Some people in HVTN 403 received an experimental HIV vaccine as a participant in a clinical trial before getting infected with HIV. Other people in this study were in a vaccine preparedness study when they got infected with HIV. None of these individuals became infected with HIV as result of their participation in an HIV vaccine or vaccine preparedness study. HVTN 403 will compare immune responses between those who previously received an experimental HIV vaccine and those who did not. Information learned from this study may be important in guiding future developments of new HIV vaccines and other treatments for HIV and AIDS.

DETAILED DESCRIPTION:
It is important to study persons vaccinated with candidate HIV-1 vaccines who have become HIV-1 infected for the following reasons. First, if transient HIV-1 infection is detected and then is effectively suppressed or cleared, it will be important to document the antigenic relationship between the breakthrough virus and the vaccine epitopes to attempt to answer questions about the specificity and breadth of the immune response and the determinants of immunity. A second reason is to gain a better understanding of vaccine-induced responses in those participants who are transiently or persistently HIV-1-infected compared to placebo recipients who become HIV-1-infected. If the vaccine does not prevent HIV-1 infection, it will be important to characterize the course of the disease as measured by longitudinal viral load measurements, CD4+ counts, and clinical symptoms. Understanding the breadth, magnitude, and specificity of the immune response in partially or fully immunized vaccinees after infection and the impact on clinical symptoms and disease progression can potentially result in valuable information for the subsequent design of vaccine efficacy trials and, ultimately, in consideration of potential effectiveness of HIV-1 vaccines.

Study visits occur at Days 0, 7, 14, 28, then at 2 months, 3 months, 6 months, and every 6 months thereafter. At these visits, patients are given a physical exam, blood is drawn, and a donation of genital fluids is requested at certain visits. Patients are asked to donate samples of either semen (men) or cervical secretions (women); viral load is measured and compared to the amount and types of virus in the blood. He/she may refuse to donate these genital fluids and still be eligible to remain in the study. Primary medical care or medications for HIV infection are not provided by this study.

ELIGIBILITY:
Inclusion Criteria

* Participated in HVTN, AVEG, HIVNET Phase I or Phase II vaccine trials or HIV vaccine preparedness trial HVTN 903 and became HIV infected after study enrollment.
* Are able and willing to provide information so that they may be located.

Exclusion Criteria

* Have a medical or mental problem that, in the opinion of the investigator, would interfere with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who were enrolled in HIV preventive vaccine clinical trials and became HIV infected as a result of the vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2002-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, Study Chair — University of Washington; Scott Hammer, MD, Study Chair — Columbia University
Locations (21):
- United States (15):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Mt Zion Hospital, San Francisco, California
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - University of MD - Inst. of Human Virology (IHV), Baltimore, Maryland
  - Jhu-Cir/Dc, Baltimore, Maryland
  - Johns Hopkins Univ, Baltimore, Maryland
  - Fenway Community Health, Boston, Massachusetts
  - Harvard University / Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Louis University School of Medicine, St Louis, Missouri
  - New York Blood Ctr / Union Square, New York, New York
  - Columbia Univ, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Miriam Hosp, Providence, Rhode Island
  - Vanderbilt Univ Hosp, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Ctr, Seattle, Washington
- Hospital Escola Sao Francisco de Assis (HESFA), Cidade Nova, Brazil
- Peru (2):
  - Asociacion Civil Selva Amazonica, Iquitos, Loreto
  - Impacta - Asociacion Civil Impacta Salud y Educaci, Lima
- South Africa (3):
  - KOSH District HVTU, Klerksdorp, North West
  - Perinatal HIV Research Unit, Chris Hani Baragwanat, Bertsham
  - University of Cape Town. Institute of Infectious Diseases, Mowbray

REFERENCES:
- [Background] Seage GR 3rd, Holte SE, Metzger D, Koblin BA, Gross M, Celum C, Marmor M, Woody G, Mayer KH, Stevens C, Judson FN, McKirnan D, Sheon A, Self S, Buchbinder SP. Are US populations appropriate for trials of human immunodeficiency virus vaccine? The HIVNET Vaccine Preparedness Study. Am J Epidemiol. 2001 Apr 1;153(7):619-27. doi: 10.1093/aje/153.7.619. PMID 11282787